CLINICAL TRIAL: NCT02273492
Title: Impact of Food on Pharmacokinetics and Pharmacodynamics of Asasantin Extended Release (ER) 200/25 mg Capsules b.i.d. in a Randomized, Open, 2-way Cross-over Study in Healthy Subjects
Brief Title: Impact of Food on Pharmacokinetics and Pharmacodynamics of Asasantin ER in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9.136
Record Dates: First submitted 2014-10-23; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (2):
- Asasantin ER after a standardized breakfast (Experimental)
  Interventions: Drug: Asasantin ER; Other: Standardized breakfast
- Asasantin ER at fasted state (Active Comparator)
  Interventions: Drug: Asasantin ER

INTERVENTIONS:
Drug: Asasantin ER
Other: Standardized breakfast
  Arms: Asasantin ER after a standardized breakfast

SUMMARY:
Comparative pharmacokinetics and pharmacodynamics of Asasantin ER at fasted and fed state

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by results of screening
* Signed written informed consent in accordance with good clinical practice (GCP) and local legislation
* Age ≥ 18 and ≤ 55 years
* Broca ≥ - 20 % and ≤ + 20 %

Exclusion Criteria:

* Any findings of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastro-intestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of hypersensitivity to Asasantin ER and any of the excipients
* Intake of drugs with a long half-life (> 24 hours) (< 1 month prior to administration or during the trial)
* Use of any drugs which might influence the results of the trial (≤ 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (< 1 month prior to administration or during the trial)
* Known alcohol abuse
* Known drug abuse
* Blood donation (< 1 month prior to administration)
* Excessive physical activities (< 5 days prior to administration)
* History of hemorrhagic diatheses
* History of gastro-intestinal ulcer, perforating or bleeding
* History of bronchial asthma
* Any laboratory value outside the normal range of clinical relevance

Female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception (adequate contraception e.g. sterilization, intrauterine devices (IUD), oral contraceptives)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 1999-08; Primary Completion 1999-10 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of dipyridamole in plasma at steady state (AUCss) | Up to 144 hours
Maximum concentration of dipyridamole in plasma at steady state (Cmax,ss) | Up to 144 hours
Change in Inhibition of cyclooxygenase for acetylsalicylic acid (ASA), analyte thromboxane B2 (TXB2) | up to day 19
Maximum concentration of dipyridamole in plasma from 0 to 10h (Cmax,0-10h) | up to 10 hours after drug administration

SECONDARY OUTCOMES:
Ratio of peak concentration of the analytes in plasma over area under the curve at steady state (Cmax,ss / AUC,ss) | Up to 144 hours
Area under the concentration-time curve of the analyte in plasma from 0 to 10 h (AUC0-10h) | Up to 10 hours after start of drug administration
Percent peak trough fluctuation of dipyridamole in plasma (%PTF) | Up to 144 hours
Time to reach the maximum concentration of the analytes in plasma at steady state (Tmax,ss) | Up to 144 hours
Terminal half-life of the analytes in plasma (t1/2) | Up to 144 hours
Percent area under the curve fluctuation of dipyridamole in plasma (AUCfluct) | Up to 144 hours
Area under the concentration-time curve of ASA in plasma at steady state (AUCss) | Up to 144 hours
Maximum concentration of ASA in plasma at steady state (Cmax,ss) | Up to 144 hours
Change in Inhibition of cyclooxygenase for acetylsalicylic acid (ASA), analyte malondialdehyde | up to day 19
Number of subjects with clinically significant changes in vital signs (blood pressure, pulse rate) | up to day 7
Number of subjects with abnormal changes in laboratory parameters | Up to 144 hours
Number of subjects with adverse events | up to 2 months